CLINICAL TRIAL: NCT00449137
Title: A Phase I Study of 5-FU (Plus Leucovorin) and Arsenic Trioxide for Patients With Refractory/Relapsed Metastatic Colorectal Carcinoma
Brief Title: Arsenic Trioxide, Fluorouracil, and Leucovorin in Treating Patients With Stage IV Colorectal Cancer That Has Relapsed or Not Responded to Treatment
Status: Completed | Phase: Phase 1 | Type: Interventional
Sponsor: University of Miami (Other)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: 20050801; SCCC-2004162
Record Dates: First submitted 2007-03-15; First posted 2007-03-19 (Estimated); Last update posted 2016-12-15 (Estimated); Status verified 2016-12

CONDITIONS: Colorectal Cancer
Keywords: recurrent colon cancer; stage IV colon cancer; recurrent rectal cancer; stage IV rectal cancer
MeSH Terms: conditions — Colorectal Neoplasms; Colonic Neoplasms; Rectal Neoplasms | interventions — Arsenic Trioxide; Fluorouracil; Leucovorin; Biopsy, Fine-Needle

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes

ARMS (1):
- Single Arm (Experimental)
  Interventions: Drug: Arsenic trioxide; Drug: Fluorouracil; Drug: Leucovorin calcium; Other: Plasma levels of elemental arsenic; Genetic: Peripheral Blood Mononuclear Cells (PBMC) for mRNA analysis; Procedure: Tumor Biopsy (Fine-Needle Aspiration)

INTERVENTIONS:
Drug: Arsenic trioxide — ATO will be administered at dose levels determined by the dose escalation scheme (section 4.2). Intra-venous (IV) infusion of ATO (mg/kg body weight) over 1-4 hours will be administered for 5 consecutive days (day 1 to day 5) during the first week, twice a week on weeks 2 and 3 (days 8, 11, 15, and 18), and only one day (day 22) of week 4. Treatment will continue for a maximum of 8 cycles, provided that the patient tolerates treatment and there is evidence of clinical benefit.
  Other Names: ATO
Drug: Fluorouracil — Escalate 5-FU, starting at dose 1600 mg/m2. On day 8, 15, and 22 the assigned dose of 5 FU plus 500 mg/m2 of leucovorin will be administered over 24 hours intravenous infusion following the administration of arsenic trioxide. Treatment will continue for a maximum of 8 cycles, provided that the patient tolerates treatment and there is evidence of clinical benefit.
  Other Names: 5-Fu
Drug: Leucovorin calcium — On day 8, 15, and 22 the assigned dose of 5 FU plus 500 mg/m2 of leucovorin will be administered over 24 hours intravenous infusion following the administration of arsenic trioxide. Treatment will continue for a maximum of 8 cycles, provided that the patient tolerates treatment and there is evidence of clinical benefit.
Other: Plasma levels of elemental arsenic — Pre-Treatment and and one hour post ATO on days 1, 5, 8, 11,15, 18, and 22
Genetic: Peripheral Blood Mononuclear Cells (PBMC) for mRNA analysis — Peripheral blood samples (PAXgene Blood RNA tube, Qiagen, USA) will be obtained up to 2 weeks prior to start of treatment (same day as the first FNA) and one hour post ATO on days 1, 5, 8, 11,15, 18, and 22. Along with FNA an additional blood sample will be obtained on day 23 of every odd treatment cycle.
Procedure: Tumor Biopsy (Fine-Needle Aspiration) — Pre-Treatment, Day 23 of Cycles 1, 3, 5, 7
  Other Names: FNA

SUMMARY:
RATIONALE: Drugs used in chemotherapy, such as fluorouracil and leucovorin, work in different ways to stop the growth of tumor cells, either by killing the cells or by stopping them from dividing. Arsenic trioxide may help fluorouracil and leucovorin work better by making tumor cells more sensitive to the drugs. Giving arsenic trioxide together with fluorouracil and leucovorin may kill more tumor cells.

PURPOSE: This phase I trial is studying the side effects and best dose of arsenic trioxide and fluorouracil when given together with leucovorin in treating patients with stage IV colorectal cancer that has relapsed or not responded to treatment.

DETAILED DESCRIPTION:
OBJECTIVES:

* Determine the maximum tolerated dose and best dose combination of fluorouracil and arsenic trioxide when given together with leucovorin calcium in patients with relapsed or refractory stage IV colorectal cancer.
* Determine if arsenic trioxide down regulates the expression of thymidylate synthase in tumor and in peripheral blood mononuclear cells in these patients.

OUTLINE: This is a dose-escalation study of fluorouracil and arsenic trioxide.

Patients receive arsenic trioxide IV over 1-4 hours on days 1-5, 8, 11, 15, 18, and 22 and fluorouracil IV over 24 hours and leucovorin calcium IV over 24 hours on days 8, 15, and 22. Treatment repeats every 5 weeks for up to 8 courses in the absence of disease progression or unacceptable toxicity.

Cohorts of 1-6 patients receive escalating doses of fluorouracil and arsenic trioxide until the maximum tolerated dose (MTD) is determined. The MTD is defined as the dose preceding that at which 2 of 3 or 2 of 6 patients experience dose-limiting toxicity. At least 6 patients are treated at the MTD.

Patients undergo peripheral blood mononuclear cell (PBMC) collection and fine-needle tumor aspiration periodically to determine the effects of arsenic trioxide on thymidylate synthase expression in the tumor and in PBMCs.

After completion of study treatment, patients are followed periodically for 3 years.

PROJECTED ACCRUAL: A total of 20 patients will be accrued for this study.

ELIGIBILITY:
DISEASE CHARACTERISTICS:

* Histologically confirmed colorectal cancer
* Stage IV disease (i.e., any T, any N, M1 disease)
* Relapsed or refractory disease

  * Disease progressed after ≥ 2 different fluorouracil-containing chemotherapy regimens (e.g., irinotecan hydrochloride or oxaliplatin with or without bevacizumab)
* Bidimensionally measurable disease
* Must have tumor amenable to biopsy and be willing to undergo fine-needle aspiration
* No CNS metastases

PATIENT CHARACTERISTICS:

* ECOG performance status 0-2
* Life expectancy > 2 months
* Platelet count > 100,000/mm^3
* WBC ≥ 3,000/mm^3
* Creatinine ≤ 1.5 times upper limit of normal
* Bilirubin ≤ 2 times normal
* SGOT ≤ 5 times normal
* Not pregnant or nursing
* Negative pregnancy test
* Fertile patients must use effective contraception during and for at least 4 months after completion of study treatment
* No preexisting peripheral neuropathy ≥ grade 2
* Ejection fraction ≥ 30%
* Baseline QT interval < 500 msec
* No serious underlying medical illness or active infection
* No underlying medical condition that could be aggravated by the treatment
* No life-threatening disease unrelated to colorectal cancer
* No other malignancy within the past 5 years unless currently disease-free and all therapy for the malignancy has been completed
* No preexisting neurological disorder (i.e., seizure disorder) ≥ grade 3
* No cardiac disease, including any of the following:

  * Recurrent supraventricular arrhythmia
  * Any type of sustained ventricular arrhythmia or conduction block (e.g., grade II or III atrioventricular block or left bundle branch block)
  * Uncontrolled ischemic heart disease
  * History of nonsustained ventricular tachycardia
  * Prolonged PR intervals (i.e., 1st degree heart block)
* No known hypersensitivity to arsenic trioxide or fluorouracil
* No history of allergic reactions attributed to compounds of similar biologic composition to arsenic trioxide or fluorouracil

PRIOR CONCURRENT THERAPY:

* See Disease Characteristics
* Recovered from all treatment-related toxicity
* At least 4 weeks since prior chemotherapy or radiotherapy and recovered
* More than 4 weeks since prior investigational drug
* No other concurrent investigational or commercial anticancer agent or therapy
* Concurrent local radiotherapy allowed for symptom relief (e.g., significant onset of pain after enrollment, but before beginning study therapy)

Ages: 18 Years to 120 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 13 (Actual)
Dates: Start 2005-06; Primary Completion 2010-02 (Actual); Study Completion 2010-12 (Actual)

PRIMARY OUTCOMES:
Maximum tolerated dose | At study completion
  The objective of this phase I study is to determine a phase II dose of combination of 5-FU and ATO that can be safely used for the treatment of 5-FU resistant colon cancer. Following the dose escalation/de-escalation procedure described in section 4.2, the recommended phase II dose of the combination 5-FU with ATO will be established as the maximum tolerated dose (MTD), defined as the highest dose level combination at which <=1 out of 6 patients experiencing DLT.
Thymidylate synthase expression | Baseline, Subsequent times
  We will characterize TS levels in study patients at baseline and at subsequent times following initiation of treatment by descriptive statistics (minimum, maximum, average, standard deviation)

CONTACTS AND LOCATIONS:
Overall Officials: Bach Ardalan, MD, Study Chair — University of Miami Sylvester Comprehensive Cancer Center
Locations (1):
- University of Miami Sylvester Comprehensive Cancer Center - Miami, Miami, Florida, United States